CLINICAL TRIAL: NCT00452088
Title: Randomized, Controlled, Dose Escalation Phase Ib Trial of MSP 3 LSP Adjuvanted in Aluminium Hydroxide Versus Hepatitis Bin 12 to 24 Month Old Children in Burkina Faso.
Brief Title: A Phase Ib Trial of MSP 3 LSP in 1-2 Year Old Children in Burkina Faso
Acronym: MSP3LSP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: African Malaria Network Trust (Network)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Dr. Roma Chilengi, African Malaria Network Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSP3_BF_0302; MSP3_BF_0302
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2007-11

CONDITIONS: Malaria
Keywords: Malaria vaccine; Safety of MSP 3 LSP; Immunogenicity of MSP 3 LSP; Burkina Faso children
MeSH Terms: conditions — Malaria | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 15 microgramme candidate vaccine group
  Interventions: Biological: MSP 3 Long Synthetic Peptide
- 2 (Active Comparator): Hepatitis B comprator group
  Interventions: Biological: Hepatitis B vaccine
- 3 (Experimental): 30 microgrammes candidate vaccine group
  Interventions: Biological: MSP 3 Long Synthetic Peptide
- 4 (Active Comparator): Hepatitis B vaccine group
  Interventions: Biological: Hepatitis B control vaccince

INTERVENTIONS:
Biological: MSP 3 Long Synthetic Peptide — Lyophilized vaccine given at 15 or 30 microgrammes
  Arms: 1; 3
Biological: Hepatitis B vaccine — Hepatitis vaccine adjuvanted in Aluminium hydroxide
  Arms: 2
Biological: Hepatitis B control vaccince — Hepatitis B vaccine adjuvanted in Aluminium hydroxide
  Arms: 4

SUMMARY:
This will be a study of the safety of MSP 3 LSP candidate malaria vaccine in children aged 1-2 years in Burkina Faso. Three imminizations at 28 day intervals will be administratered subcuteneously on the shoulder region. The study will compare MSP3 with Engerix B vaccine to evaluate whether it is just as safe to give to children in malaria endemic country. The study will also evaluate whether the vaccine induces the expected immune responses. Two dose levels of MSP 3 will be evaluated; 15µg and 30µg to determine the one with the best safety and immune response profile.

DETAILED DESCRIPTION:
The study is a single centre randomized controlled and blinded study (observer blind). It will be conducted at the CNRFP Vaccinology unit located in Balonghin. Children in the catchments area within the 1-2 years age group, whose parents consent will be screened to randomise 45 eligible participants. Two MSP 3 dose levels will be evaluated; 15µg and 30µg. The study will start with immunizing older children with the lowest dose observing safety parameters closely, then proceed to to the higher dose with a two week of observation apart.

Clinical, biological and immune response data gathered after vaccination with 15µg and 30µg MSP 3 LSP will be compared to:

* The children's baseline data before vaccinations, and
* The post vaccination data of children in the control group.

Randomization will ensure that the comparison groups are similar in relevant characteristics at baseline. The concealment of allocation before enrolment will further enforce the randomisation. Individuals who will make the assessment of the study end points will be completely blinded of the vaccine administered. This will ensure that there is no observer bias. Further, reporting or information bias will be minimised, because the recipients will also not be aware of which vaccine they have been administered. This is possible because the selected control vaccine has not been in routine use in this area, and has only now been recommended by the Ministry of Health. Cross over immunisation at the end of the trial will involve only those children who will received the study vaccine; they will be administered the control vaccine in the interest of public health benefits for them.

The schedule of vaccination at 0, 1 and 2 months has been adopted because it is suitable for the target group. The idea is to eventually deploy the vaccine through the expanded programme on immunisation should the vaccine become registered for public use. For the EPI age group, it is not only an efficient delivery mechanism, but they are also the most vulnerable group to malaria.

In brief, the groups will be allocated as follows:

* Group 1: 23 participants (15 receiving MSP-3 vaccine 15 µg and 8 receiving Hepatitis B vaccine).
* Group 2: 22 participants (15 receiving MSP-3 vaccine 30 µg and 7 receiving Hepatitis B vaccine)

Immunization schedule will be 0, 1, and 2 months for all cohorts and provisionally as following for each group:

Study days 0, 28 and 56 for group 1; and Study days 14, 42, 70 for group 2 Vaccinations of groups 1 and 2 will be staggered: immunization in group 2 will start 2 weeks after group 1. This interval may be extended if deemed necessary due to SAEs or other safety concerns.Randomization will be done for each group at the times of first vaccinations.Route of inoculation will be by subcutaneous injection into right or left deltoid (alternately).

Each child will be observed for at least 60 minutes after vaccination to evaluate and treat any acute adverse events (AEs). Study duration will be approximately 13 months per participant. There will be a seven (7) day follow-up period for solicited adverse events (day of vaccination plus 6 subsequent days); and twenty eight (28) day follow-up period for unsolicited adverse events (Vaccination day plus 27 subsequent days). The follow-up for serious adverse events (SAE's) will be for 12 months following the first dose of study vaccine (9 months after dose 3).

At the end of the follow-up period for unsolicited AEs (i.e., one month after the third dose), participants will be followed by field workers at home at monthly intervals to record SAEs. For data collection, conventional paper Case Report Forms (in triplicate copies) will be used.

An interim analysis is foreseen after day 84 of follow up. At this stage decision will be considered whether to proceed to a phase 2b study or not, and with which dosage of MSP 3, based on the safety and immunogenicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-2 years old
* Healthy by medical history and physical examination
* Signed Informed Consent by guardian/parent
* Resident in the study area village during the whole trial period

Exclusion Criteria:

* Symptoms, physical signs of disease that could interfere with the interpretation of the trial results or compromising the health of the subjects
* Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior recruitment. (for corticosteroids, this will mean prednisone, or equivalent,0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Cannot be followed for any social, psychological or geographical reasons.
* Use of any investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose.
* Suspected or known hypersensitivity to any of the vaccine components or to previous vaccine.
* Laboratory abnormalities on screened blood samples out of range, more specifically refer to table 2.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine. An exception, is the receipt of an EPI or licensed vaccine (measles, oral polio, Hib, meningococcal and combined diphtheria, pertussis,tetanus vaccines) which may be given 14 days or more before or after vaccination
* Evidence of chronic or active hepatitis B infection
* Presence of chronic illness that, in the judgement of the investigator, would interfere with the study outcomes or pose a threat to the participant's health.
* Administration of immunoglobulin andor any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* History of surgical splenectomy.
* Moderate or severe malnutrition at screening defined as weight for age Z score less than 2

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Immediate reactogenicity (within 1 hour, with emphasis on allergic reactions) | 7 days
Local and systemic reactogenicity during the 7 days following the vaccine | 7 days
Unsolicited adverse events occurring within 28 days following each vaccination | 28 Days
Serious adverse events (SAE) throughout the study period | 1 year

SECONDARY OUTCOMES:
Humoral immune responses by ELISA before and four weeks after each vaccination | 84 Days
Cellular immune response to the vaccine antigens by measuring the | 84 Days
number of cells producing IFNγ/106 cells by Elispot to MSP3-LSP and | 84 Days

CONTACTS AND LOCATIONS:
Overall Officials: Issa Nebie, PhD, Study Director — Projet de Développement de Vaccins Anti-Paludique- Centre National de Recherche et de Formation sur le Paludisme
Locations (1):
- Projet de Développement de Vaccins Anti-Paludique- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Sapone, Burkina Faso

REFERENCES:
- [Derived] Sirima SB, Tiono AB, Ouedraogo A, Diarra A, Ouedraogo AL, Yaro JB, Ouedraogo E, Gansane A, Bougouma EC, Konate AT, Kabore Y, Traore A, Chilengi R, Soulama I, Luty AJ, Druilhe P, Cousens S, Nebie I. Safety and immunogenicity of the malaria vaccine candidate MSP3 long synthetic peptide in 12-24 months-old Burkinabe children. PLoS One. 2009 Oct 26;4(10):e7549. doi: 10.1371/journal.pone.0007549. PMID 19855847